Informed Consent Hopewell Hospitalist: A Video Game Intervention to Increase Advance Care Planning by Hospitalists [Efficacy Trial]

NCT 04557930 11 March 2020

### **Dartmouth College**

Study Title: Video Games for Clinician Decision-Making: Efficacy

Principal Investigator: Amber E. Barnato MD MPH MS

You are being asked to take part in a research study. Taking part in research is voluntary.

Thank you for your willingness to participate in this study. This study is part of an NIH-funded research project about how clinicians make decisions. The study will take **approximately 3 hours to complete.** 

### Participation:

Your participation is entirely voluntary. Refusal to participate, withdrawal of your consent, or discontinued participation in the study will not result in any penalty or loss of benefits to which you might otherwise be entitled.

We will provide you with an iPad for participating in this study. This is for your time and personal cost of participation.

## What this study involves:

You will be asked to play an interactive video game for approximately 3 hours over the course of 2 weeks. Before and after the game, you will be asked to complete short questionnaires. This will include questions about your general background and your experiences with the game. Your responses will also be linked to Sound billing or other Medicare claims data.

# Risks:

The primary risk associated with this study is loss of confidentiality. Other risks and discomfort associated with participation in this study are no greater than those ordinarily encountered in daily life.

Your identity will be kept confidential and maintained during data analysis and publication/presentation of results by the following means: (1) Your responses to the survey will be electronically anonymized after being linked to Sound billing or other Medicare claims data; (2) The researchers will store the data file by your number, not by name. (3) Only members of the research group will view collected data in detail. (4) Any files will be stored in a secured location accessed only by authorized researchers. (5) No identifiable information will be reported to your employer, including whether or not you complete study procedures.

#### **Questions and Contacts**

If you have any questions about this study, you should feel free to ask them now or anytime throughout the study by contacting:

Amber E. Barnato MD MPH MS
The Dartmouth Institute for Health Policy & Clinical Practice

1 Medical Center Dr, Lebanon, NH 03766 Email: <a href="mailto:amber.barnato@dartmouth.edu">amber.barnato@dartmouth.edu</a>

Phone: 603-653-0829

1

If you have questions pertaining to your rights as a research participant; or to report objections to this study, you should contact:

Committee for the Protection of Human Subjects 63 South Main Street, Room 302 Hanover, NH 03755

Phone: (603) 646-6482 Fax: (603) 646-9141

Email: cphs@dartmouth.edu

# **CONSENT**

I understand the nature of this study and agree to participate. I received a copy of my consent. I give the Principal Investigator, and his/her associates, permission to present this work in written and/or oral form for teaching or presentations to advance the knowledge of science and/or academia, without further permission from me provided that my image or identity is not disclosed.

I have read the above information about *Video Games for Clinician Decision-Making* and have been given time to ask questions. I agree to take part in this study and I will be given a copy of this signed consent form.

Click to agree to participate